CLINICAL TRIAL: NCT04757519
Title: Enhancing the Diabetes Prevention Program to Promote Weight Loss Among Nonresponders in a Community-Based Lifestyle Intervention.
Brief Title: Enhanced DPP-GLB to Promote Weight Loss Among Nonresponders in a Community-Based Lifestyle Intervention.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lovoria Williams (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Lovoria Williams, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 58766; 1R01DK125801-01 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-02-17 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Diabetes
Keywords: prevention; weight loss; community; personalized; telephone; resources; lifestyle intervention; racial ethnic minorities / African American; faith based; obesity; non-responders; adults; cancer
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss; Obesity; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPP-GLB Standard (Experimental): Participants in this group will receive the standard Diabetes Prevention Program Group Lifestyle Balance (DPP-GLP) Intervention Program.
  Interventions: Behavioral: DPP-GLB Standard
- DPP-GLB Enhanced (Experimental): Participants in this group will receive the enhanced Diabetes Prevention Program Group Lifestyle Balance (DPP-GLP) Intervention Program.
  Interventions: Behavioral: DPP-GLB Enhanced

INTERVENTIONS:
Behavioral: DPP-GLB Standard — The intervention is based upon the 2017 version of the University of Pittsburgh DPP Group Lifestyle Balance Program (DPP-GLB). Participants will receive the DPP-GLB intervention once per week for 12 weeks, then twice monthly for 12 weeks (18 sessions total). The program includes hour-long group-based sessions and supportive materials including a weekly food diary and FitBit/pedometer.
  Arms: DPP-GLB Standard
Behavioral: DPP-GLB Enhanced — The intervention is based upon the 2017 version of the University of Pittsburgh DPP Group Lifestyle Balance Program (DPP-GLB). Participants will receive the DPP-GLB intervention once per week for 12 weeks, then twice monthly for 12 weeks (18 sessions total). The program includes hour-long group-based sessions and supportive materials including a weekly food diary and FitBit/pedometer. Intervention week 4, weight loss non-responders defined as weight loss less than 1% receive weekly telephone intervention, using motivational interviewing techniques to provide social support, assess barriers, resolve ambivalence, and support the participant in developing personal strategies. Additionally, this intervention includes weekly phone calls using motivational interviewing techniques to provide social support, assess barriers, resolve ambivalence, and support the participant in developing personal strategies. Links to relevant videos may also be provided.
  Arms: DPP-GLB Enhanced

SUMMARY:
This study seeks to establish the efficacy of identifying weight loss nonresponders early in a Diabetes Prevention Program (DPP) intervention in 20 community settings (primarily churches and community centers) and providing them with individual-level, enhanced treatment through telephone contacts and access to additional resources. Additionally, potential mediators and moderators of the relationship between intervention status and weight loss response at 6 months in both nonresponders and responders will be examined and a cost-effectiveness analysis to evaluate the cost of the intervention will be conducted.

This study addresses key gaps in the literature about the weight loss effects of identifying nonresponders early and characterizing individuals who need more intense personalized strategies. The investigators hypothesize that changes between baseline and 3 months will be more pronounced among the nonresponders in the intervention group compared to the nonresponders in the active control group.

ELIGIBILITY:
Inclusion Criteria:

* self-described as Black
* non-diabetic
* body mass index (BMI) equal to or greater than 25
* CDC diabetes risk assessment greater than or equal to 5 or diabetes pre-diagnosis or history of gestational diabetes
* live within driving distance of participating church/site

Exclusion Criteria:

* diagnosed Type 1 or 2 diabetes
* pregnant or planning to become pregnant during study period
* contraindications to moderate physical activity
* serious medical condition that contradicts weight loss
* not Black or African American

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lovoria Williams, Principal Investigator — University of Kentucky
Locations (21):
- United States (21):
  - First Corinthian Baptist Church, Frankfort, Kentucky
  - Heavenly Outpour, Frankfort, Kentucky
  - Consolidated Baptist Church, Lexington, Kentucky
  - Historic St. Paul AME Church, Lexington, Kentucky
  - First African Baptist Church, Lexington, Kentucky
  - Pilgrim Baptist Church, Lexington, Kentucky
  - Shiloh Baptist Church, Lexington, Kentucky
  - Redeemed Christian Church of God, Lexington, Kentucky
  - First Baptist Church Brackstown, Lexington, Kentucky
  - Lima Drive Seventh Day Adventist Church, Lexington, Kentucky
  - Kingdom Fellowship, Louisville, Kentucky
  - Bates Memorial Baptist Church, Louisville, Kentucky
  - St. Stephen Baptist Church, Louisville, Kentucky
  - Greater Gaililee CDC, Louisville, Kentucky
  - Historic Calvary MBC, Louisville, Kentucky
  - Spirit Filled New Life Church, Louisville, Kentucky
  - Forest Baptist Church, Louisville, Kentucky
  - Burnett Ave BC, Louisville, Kentucky
  - Marnel C. Moorman Family Life Center, Shelbyville, Kentucky
  - New Mt. Zion Baptist Church, Shelbyville, Kentucky
  - First Baptist Winchester, Winchester, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams LB, Moser DK, Gustafson A, Waters TM, Rayens MK, Karle ER, Kriska AM. Reaching high-risk Black adults for diabetes prevention programming during a pandemic: The design of Fit & Faithful a randomized controlled community trial. Contemp Clin Trials. 2022 Dec;123:106973. doi: 10.1016/j.cct.2022.106973. Epub 2022 Nov 5. PMID 36334705

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Churches
Period: Overall Study
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Started | 203; 10 Churches | 200; 10 Churches
Completed | 186; 10 Churches | 182; 10 Churches
Not Completed | 17; 0 Churches | 18; 0 Churches
Not completed — Lost to Follow-up | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced | Total
Number analyzed (Participants) | 203 | 200 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed in the row differs from the overall due to some participants consenting and enrolling, but withdrawing before the first data collection.
  years
    number analyzed (Participants) | 186 | 182 | 368
    (all) | 55.9 (12.2) | 53.2 (12.1) | 54.56 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed in the row differs from the overall due to some participants consenting and enrolling, but withdrawing before the first data collection.
  Participants
    number analyzed (Participants) | 186 | 182 | 368
    Female | 158 | 163 | 321
    Male | 28 | 19 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American / Black | 203 | 200 | 403
Region of Enrollment [Number; unit: participants]
  United States | 203 | 200 | 403
Married/partnered [Count of Participants; unit: Participants] | 87 | 86 | 173
College or graduate degree [Count of Participants; unit: Participants] | 109 | 106 | 215
Private Insurance [Count of Participants; unit: Participants] | 120 | 120 | 240
Income > $50,000 annually [Count of Participants; unit: Participants] | 93 | 95 | 188

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight at 12 Weeks
Description: Weight will be measured in pounds using a cellular scale at baseline and at 12 weeks.
Time Frame: 12 weeks (at baseline and12 weeks)
Population: Participants who completed the 12-week data collection.
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 176 | 168
pounds (lbs)
  Baseline | 230.48 (52.22) | 225.94 (46.24)
  12-Week | 224.71 (51.3) | 219.30 (44.51)

2. Primary Outcome: Change in Weight at 6 Months
Description: Weight will be measured in pounds using a cellular scale at baseline and at 6 months.
Time Frame: 6 months (at baseline and 6 months)
Population: Participants who completed the 6-month data collection.
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 167 | 165
pounds (lbs)
  Baseline | 230.48 (52.22) | 225.94 (46.24)
  6-Month | 223.16 (51.8) | 216.44 (44.31)

3. Secondary Outcome: Change in Blood Pressure at 12 Weeks
Description: Blood pressure will be measured with calibrated automated blood pressure monitor at baseline and at 12 weeks.
Time Frame: 12 weeks (at baseline and 12 weeks)
Population: Participants who completed the 12-week data collection.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm Hg)
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 173 | 165
Millimeters of mercury (mm Hg)
  Baseline Systolic | 138 (16) | 138 (17)
  Baseline Diastolic | 78 (10) | 80 (11)
  12 Weeks Systolic | 133 (14) | 136 (15)
  12 Weeks Diastolic | 77 (10) | 79 (11)

4. Secondary Outcome: Change in Blood Pressure at 6 Months
Description: Blood pressure will be measured with calibrated automated blood pressure monitor at baseline and at 6 months.
Time Frame: 6 months (at baseline and 6 months)
Population: Those who participated in 6-month data collection.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm Hg)
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 167 | 161
Millimeters of mercury (mm Hg)
  Baseline Systolic | 138 (16) | 138 (17)
  Baseline Diastolic | 78 (10) | 80 (11)
  6 Month Systolic | 135 (17) | 134 (15)
  6 Month Diastolic | 78 (12) | 78 (11)

5. Secondary Outcome: Change in Physical Activity at 12 Weeks
Description: Change in Physical Activity will be measured at baseline and 12-week using the Modifiable Activity Questionnaire (MAQ), which assesses activity frequency and duration across the leisure and occupational components. Responses were converted to metabolic equivalent hours per week (MET-hrs/week) using standard scoring procedures, where higher MET-hrs/week indicates greater physical activity.
Time Frame: 12 weeks (at baseline and 12 weeks)
Population: Participants who completed 12-week data collection and said yes to performing any form of physical activity listed on the MAQ
Measure: Mean (Standard Deviation); unit: MET-hrs/week
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 158 | 151
MET-hrs/week
  Baseline | 9.2 (10) | 6.5 (7.4)
  12 Weeks | 13.8 (12.8) | 12.2 (13.6)

6. Secondary Outcome: Change in Physical Activity at 6 Months
Description: Change in Physical Activity will be measured at baseline and 6-month using the Modifiable Activity Questionnaire (MAQ), which assesses activity frequency and duration across the leisure and occupational components. Responses were converted to metabolic equivalent hours per week (MET-hrs/week) using standard scoring procedures, where higher MET-hrs/week indicates greater physical activity.
Time Frame: 6 months (at baseline and 6 months)
Population: Participants who completed 6-month data collection and said Yes to performing a form of activity on MAQ.
Measure: Mean (Standard Deviation); unit: MET-hrs/week
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 144 | 123
MET-hrs/week
  Baseline | 9.2 (10) | 6.5 (7.4)
  6 Months | 14.47 (13.02) | 10.49 (9.69)

7. Secondary Outcome: Change in Dietary Intake at 12 Weeks
Description: Change in Dietary Intake will be measured using the validated, Dana Farber eating habits tool and the Dietary screener questionnaire which assesses the frequency of consumption of selected foods and drinks. The scoring range of the survey is Never or less than once per month, 1-3 per month, 1 per week, 2-4 per week, 5-6 per week, 1 per day, 2-3 per day, 4-5 per day, 6 or more per day, Prefer not to answer. Higher scores indicated increased dietary intake. The total score is the sum of the scores on all items, divided by the total maximum score possible, and then multiplied by 100.
Time Frame: 12 weeks (at baseline and 12 weeks)
Population: Participants who completed the 12-week data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 167 | 152
score on a scale
  Baseline | 69.86 (14.22) | 68.13 (14.22)
  12 Weeks | 72.22 (13.22) | 71.52 (13.15)

8. Secondary Outcome: Change in Dietary Intake at 6 Months
Description: Change in Dietary Intake will be measured using the validated, Dana Farber eating habits tool and the Dietary screener questionnaire which assesses the frequency of consumption of selected foods and drinks. The scoring range of the survey is Never or less than once per month, 1-3 per month, 1 per week, 2-4 per week, 5-6 per week, 1 per day, 2-3 per day, 4-5 per day, 6 or more per day, Prefer not to answer. Higher scores indicated increased dietary intake.The total score is the sum of the scores on all items, divided by the total maximum score possible, and then multiplied by 100.
Time Frame: 6 months (at baseline, 12 weeks, 6 months)
Population: Those who participated in 6-month data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 160 | 156
score on a scale
  Baseline | 69.86 (14.22) | 68.13 (14.22)
  6 Month | 71.11 (15.0) | 70.08 (13.15)

9. Secondary Outcome: Cost Analysis
Description: Investigator-developed instrument. At 6 months, conduct a cost-effectiveness analysis to evaluate the cost of the intervention arm by comparing the incremental cost and weight loss with the active control arm. The generated final output is the cost per participant in dollars.
Time Frame: 6 months
Population: Participants who completed the 6-month data collection.
Measure: Mean (Standard Deviation); unit: dollar
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 186 | 182
dollar | 471.49 (75.25) | 461.06 (39.87)

10. Secondary Outcome: Impact of Weight on Quality of Life
Description: Quality of life will be measured using Impact of Weight on Quality of Life Questionnaire (IWQOL-Lite). This is a 31-item self-report scale. Scores range from 0-100; higher scores indicate greater quality of life.
Time Frame: 6 months
Population: Participants who completed the 6-month data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
Number analyzed (Participants) | 141 | 148
score on a scale | 44.75 (16.66) | 47.10 (18.15)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DPP-GLB Standard | DPP-GLB Enhanced
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/200
Other Adverse Events (participants affected / at risk) | 0/203 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT04757519/Prot_SAP_001.pdf
  • Informed Consent Form (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04757519/ICF_000.pdf